CLINICAL TRIAL: NCT04274790
Title: Analysis of the Impact of 5-Fluorouracil on the Translational Control and Plasticity of Cancer Cells From Liver Metastases of Colon Cancer
Brief Title: Impact of 5-Fluorouracil (5-FU) on Cancer Cells From Liver Metastases of Colon Cancer
Acronym: FLUORIB
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET 19-127 FLUORIB
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Colon; Metastasis to Liver
MeSH Terms: conditions — Colonic Neoplasms | interventions — Appointments and Schedules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A fragment of the previously operated primary tumor: block and/or archived frozen tumor if available.
  * A fragment of the liver metastasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic colon cancer: Patient with metastatic colon cancer operated on and followed up at the Centre Leon Berard for liver metastasis.
  Interventions: Procedure: Scheduled and planned surgery

INTERVENTIONS:
Procedure: Scheduled and planned surgery — Collection of tumour samples from samples collected as part of standard patient management. Diagnostic pathological analysis will be a priority. These samples will be taken by experienced staff during the hospital visit scheduled as part of standard care.

SUMMARY:
Analyze the dynamics of incorporation of 5-fluorouracil into cancer cell ribosomes from liver metastases of patient with metastatic colon cancer.

DETAILED DESCRIPTION:
This is a monocentric, prospective, non-interventional cohort study in adult patients with metastatic colon cancer with hepatics metastasis.

Tumour samples collected for this study include:

* A fragment of the previously operated primary tumor: FFIP block and/or archived frozen tumor if available.
* A fragment of the liver metastasis(s) performed as part of standard metastasis surgery, this fragment will include a tumor area and a healthy area within the margin of excision. These samples collected in a fresh state will be analyzed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic colon cancer operated on and followed up at the Centre Leon Berard for liver metastasis.
* Patient affiliated to social security

Exclusion Criteria:

* Other pathologies that may interfere with biological evaluation, in particular known hepatic cirrhosis, whatever its origin, other liver overload diseases (hemochromatosis, Wilson's disease), but excluding steatosis (which can be chemo-induced).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic colon cancer in the hepatic phase.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
5-FU in ribosome | Up to 24 months
  Rate of incorporation of 5-fluorouracil into ribosomes of tumor tissues and adjacent healthy tissues before surgery and after surgery.

SECONDARY OUTCOMES:
Methylation profile of ribosomal RNAs | Up to 24 months
  Analyze on a large scale the alterations of the 2'-O-methylation profile of ribosomal RNAs before surgery and after surgery
Transcriptomic and proteomic profile | Up to 24 months
  Define a transcriptomic and proteomic profile of the collected samples before surgery and after surgery.
Specific molecular signature | Up to 24 months
  Combination of the number of 5-fluorouracil molecules incorporated per rRNA molecule, the methylation profile and the transcriptomic profile before surgery and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France